CLINICAL TRIAL: NCT06624592
Title: Sevoflurane/Dexmedetomidine vs. Isoflurane and Their Effects on Pediatric Emergence Delirium
Brief Title: Sevoflurane/Dexmedetomidine vs. Isoflurane for Pediatric Emergence Delirium
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Lindsay L. Warner, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-002252
Record Dates: First submitted 2024-08-21; First posted 2024-10-03 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Delirium on Emergence
MeSH Terms: conditions — Emergence Delirium | interventions — Sevoflurane; Isoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Isoflurane group (Active Comparator)
  Interventions: Drug: Isoflurane
- Sevoflurane group (Active Comparator)
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — Subjects will receive standard of care anesthesia Sevoflurane, with intravenous push Dexmedetomidine
  Arms: Sevoflurane group
Drug: Isoflurane — Subjects will receive standard of care anesthesia Isoflurane
  Arms: Isoflurane group

SUMMARY:
The purpose of this study is to measure the incidences of pediatric emergence delirium between the group receiving Isoflurane and the group receiving Sevoflurane plus intravenous push dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 2-7 years.
* Surgeries include ENT cases (i.e., tonsillectomy/adenoidectomy), ophthalmology cases (i.e., strabismus), and urology cases.
* Can be outpatient or General Care inpatient procedures.
* All cases must include an IV and an endotracheal tube (ETT).

Exclusion Criteria:

* Severe developmental/cognitive delay (unable to make eye contact, nonverbal, or inability to interact with providers for PAED scale assessment requirements)
* TIVA cases.
* No PIV in place during the case, planned PICU admission postoperatively.
* Previous history of severe emergence delirium documented by a provider (via interventions or explicitly stated).

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with emergence delirium | Within 1 hour after dropped off by anesthesiology team
  Total number of subjects with a Pediatric Anesthesia Emergence Delirium (PAED) score of > 10. The PAED scale consists of 5 criteria that are scored using a 5-point scale. The scores of each criterion are added to make a total score. The maximum achievable total score is 20.

SECONDARY OUTCOMES:
Post Anesthesia Care Unit (PACU) length of stay | Post-procedural (0-4 hours after anesthesiology drop off)
  Number of hours spent in PACU during recovery

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Warner, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No